CLINICAL TRIAL: NCT02887508
Title: Internet-based STI/HIV Prevention for HIV+ Internet Users
Brief Title: HIV Internet Sex Study: Internet-based STI/HIV Prevention for HIV+ Internet Users
Acronym: HINTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dean Cruess, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H10-217; R34MH087120 (NIH)
Record Dates: First submitted 2016-08-24; First posted 2016-09-02 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: HIV-1 Infection; Risk Reduction
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HINTS Intervention (Experimental): The HINTS intervention consisted of an online four-session group intervention for 45 minutes, twice a week for two weeks. In each session, facilitators presented information, motivational skills, and behavioral skills related to a specific topic relevant to online partner seeking and transmission risk reduction, including Internet safety and communication, condom negotiation, and serostatus disclosure.
  Interventions: Behavioral: HINTS Intervention
- Healthy Living Control (Active Comparator): The Healthy Living Control condition consisted of an online four-session group intervention for 45 minutes, twice a week for two weeks. In each session, facilitators presented information, motivational skills, and behavioral skills to address non-sexual health-related topics particularly relevant to individuals living with HIV, such as nutrition, healthy eating, portion control, exercise and staying active, and stress reduction.
  Interventions: Behavioral: Healthy Living Control

INTERVENTIONS:
Behavioral: HINTS Intervention — HINTS is a four-session, group-based behavioral intervention delivered exclusively online and developed using the IMB model of health behavior change focused on sexual risk reduction.
  Arms: HINTS Intervention
Behavioral: Healthy Living Control — The Healthy Living Control is a four-session, group-based behavioral intervention delivered exclusively online and developed using the IMB model of health behavior change focused on non-sexual health topics.
  Arms: Healthy Living Control

SUMMARY:
The goal of this study was to empirically test a newly developed online HIV sexual risk reduction intervention (HINTS) among a representative sample of gay and bisexual men living with HIV who meet sex partners online.

DETAILED DESCRIPTION:
Internet-based venues such as websites, chat rooms, blogs, and bulletin boards are becoming an increasingly popular means for HIV-positive men who have sex with men (MSM) to meet potential sex partners. The anonymity, quickness, and convenience offered by online venues allows for numerous potential sex partners to be identified and screened with the possibility to meet in person. However, there are potential health hazards associated with meeting sex partners online, including an increased risk of sexually transmitted infections (STIs), and thus there is an urgent need for online behavioral interventions to help reduce STI/HIV risks associated with Internet-initiated sexual liaisons. This research involves developmental intervention studies to design and field test an online, theory-based behavioral risk reduction intervention for HIV-positive MSM who use the Internet to meet potential sex partners. Guided by the Information-Motivation-Behavioral Skills (IMB) model of health promoting behaviors the investigators will conduct 3 stages of intervention development research, as follows: (1) perform initial interviews and focus groups with HIV-positive MSM who use the Internet to meet sex partners. Stage 1 will also bring together expert and community consultants to aid in the intervention development. Based on information gained from rapid formative studies, this first stage of research will directly lead to the development a novel online theory-based sexual risk reduction intervention; (2) test the feasibility and acceptability of the newly developed online STI/HIV risk reduction intervention with a sample of HIV-positive MSM who use the Internet to meet sexual partners. Stage 2 will also involve programming an audio-computer assisted interview for data collection; and (3) conduct a randomized field test to determine the potential efficacy of the risk reduction intervention for MSM who use the Internet to potentially meet sex partners. Participants in the field test will be randomly assigned to either receive the newly developed intervention or a time-matched attention comparison condition. Stage 3 will include testing for differences between groups on behavioral risk and Internet use outcomes across a 6-month follow-up period. The investigators will also examine the intervention effects on mediating and moderating constructs of information, motivation, and behavioral skills. The proposed intervention research will therefore develop new STI/HIV prevention strategies delivered exclusively online for use with people living with HIV/AIDS (PLWHA) who use the Internet to meet potential sex partners. The results from this study will provide preliminary data on which to conduct a larger-scale, randomized controlled clinical trial in the future.

ELIGIBILITY:
Inclusion Criteria:

1. being over 18 years of age
2. self-identifying as gay or bisexual
3. living with HIV/AIDS
4. reporting having used the Internet at least once to meet a potential sex partner
5. reporting any history of unprotected anal sex with a male partner.

Exclusion Criteria:

1. non-fluency in English
2. inability to participate in online group intervention

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2010-12; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Sexual risk behavior, such as condomless anal sex with sexual partners, will be assessed via a self-report survey. Data will be aggregated and reported as counts or occurrences. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dean G Cruess, PhD, Principal Investigator — University of Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Burnham KE, Cruess DG, Kalichman MO, Grebler T, Cherry C, Kalichman SC. Trauma symptoms, internalized stigma, social support, and sexual risk behavior among HIV-positive gay and bisexual MSM who have sought sex partners online. AIDS Care. 2016;28(3):347-53. doi: 10.1080/09540121.2015.1096894. Epub 2015 Oct 13. PMID 26461452
- See also: Baseline manuscript — http://www.ncbi.nlm.nih.gov/pubmed/26461452